CLINICAL TRIAL: NCT03532880
Title: A Phase I Study of Olaparib and Low Dose Thoracic Radiotherapy for Extensive Stage Small Cell Lung Cancer
Brief Title: A Study of Olaparib and Low Dose Radiotherapy for Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-195
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Carcinoma
Keywords: Olaparib; Radiation therapy; 18-195; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — olaparib; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Small Cell Lung Cancer (Experimental)
  Interventions: Drug: Olaparib Pill 50 mg; Drug: Olaparib Pill 100 mg; Drug: Olaparib Pill 150 mg; Drug: Olaparib Pill 200 mg; Drug: Olaparib Pill 250 mg; Drug: Olaparib Pill 300 mg; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Olaparib Pill 50 mg — Olaparib dosing will be twice-daily (BID) dosing. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Drug administration at the dose level will occur on Day 1 (6 - 9 days prior to start of radiotherapy; for logistical considerations this may occur on the day of simulation for radiotherapy) and will continue concurrently with low dose consolidative thoracic radiotherapy until last day of radiotherapy (Day 20 - 23)
Drug: Olaparib Pill 100 mg — Olaparib dosing will be twice-daily (BID) dosing. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Drug administration at the dose level will occur on Day 1 (6 - 9 days prior to start of radiotherapy; for logistical considerations this may occur on the day of simulation for radiotherapy) and will continue concurrently with low dose consolidative thoracic radiotherapy until last day of radiotherapy (Day 20 - 23)
Drug: Olaparib Pill 150 mg — Olaparib dosing will be twice-daily (BID) dosing. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Drug administration at the dose level will occur on Day 1 (6 - 9 days prior to start of radiotherapy; for logistical considerations this may occur on the day of simulation for radiotherapy) and will continue concurrently with low dose consolidative thoracic radiotherapy until last day of radiotherapy (Day 20 - 23)
Drug: Olaparib Pill 200 mg — Olaparib dosing will be twice-daily (BID) dosing. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Drug administration at the dose level will occur on Day 1 (6 - 9 days prior to start of radiotherapy; for logistical considerations this may occur on the day of simulation for radiotherapy) and will continue concurrently with low dose consolidative thoracic radiotherapy until last day of radiotherapy (Day 20 - 23)
Drug: Olaparib Pill 250 mg — Olaparib dosing will be twice-daily (BID) dosing. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Drug administration at the dose level will occur on Day 1 (6 - 9 days prior to start of radiotherapy; for logistical considerations this may occur on the day of simulation for radiotherapy) and will continue concurrently with low dose consolidative thoracic radiotherapy until last day of radiotherapy (Day 20 - 23)
Drug: Olaparib Pill 300 mg — Olaparib dosing will be twice-daily (BID) dosing. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water.
  Drug administration at the dose level will occur on Day 1 (6 - 9 days prior to start of radiotherapy; for logistical considerations this may occur on the day of simulation for radiotherapy) and will continue concurrently with low dose consolidative thoracic radiotherapy until last day of radiotherapy (Day 20 - 23)
Radiation: Radiotherapy — The total prescribed dose will be 30 Gy in ten daily fractions of 3 Gy each delivered during business days over 2 calendar weeks.

SUMMARY:
The purpose of this study is to test the safety of a new medication, Olaparib, combined with radiation therapy for participants with small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological documented diagnosis of SCLC confirmed by a MSKCC pathologist.
* Documented extensive disease, defined as any tumor beyond the above limited disease definition, including ipsilateral lung metastases and malignant pleural effusion
* Completion of induction chemotherapy with a minimum of 4 and no more than 6 cycles of a platinum agent and etoposide within 8 weeks of trial initiation.
* No disease progression (i.e.SD or better response per treating physician descretion) at the completion of chemotherapy.
* Age 18 years or older.
* Intrathoracic disease should be encompassable in acceptable radiation fields per investigator clinical judgement.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnosfsky Performance Score (KPS) >/= 70
* Patients must have adequately recovered from any adverse events associated with prior immune-chemotherapy
* Adequate organ and marrow function, including:

  1. Haemoglobin >/= 8.0 g/dL with no blood transfusion in the past 28 days.
  2. Absolute neutrophil count (ANC) >/= 1.5 x 10^9/L.
  3. Platelet count >/= 100 x 10^9/L.
  4. Total bilirubin </= 1.5 x institutional upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) </= 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be </= 5x ULN.
  6. Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of >/= 51 mL/min
* Patients must have a life expectancy >/= 16 weeks.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

  a. Postmenopausal is defined as any one or more of the following: i. Age >/= 60 years. ii. Age < 60 and amenorrheic for 1 year or more in the absence of chemotherapy and/or hormonal treatment.

iii. Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 60.

iv. Radiation-induced oophorectomy with last menses >1 year ago v. Chemotherapy-induced menopause with > 1 year interval since last menses. vi. Surgical sterilisation (bilateral oophorectomy or hysterectomy).

* Men and women of childbearing potential must be willing to us two highly effective forms of contraception while on treatment and for at least 3 months after last dose of study drug.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Written informed consent

Exclusion Criteria:

* Untreated brain metastases.
* Pneumonitis
* Previous radiotherapy to thorax (prior breast RT is permitted).
* Patient is not a candidate for or declines consolidative thoracic radiotherapy.
* Patients receiving any systemic chemotherapy or thoracic radiotherapy within 3 weeks prior to study treatment.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Previous enrolment in the present study.
* Exposure to an investigational product within 30 days or 5 half lives (whichever is longer) prior to start of the current study drug.
* Any previous treatment with PARP inhibitor, including olaparib, for the treatment of small cell lung cancer
* Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or a documented family history of long QT syndrome.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong CYP3A inducers (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* For patients who have received prior immunotherapy, treatment must be held from 10 days prior to protocol treatment until 10 days after completing protocol treatment.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome/acute leukaemia or with features suggestive thereof.
* Major surgery within 2 weeks of study treatment initiation and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active/uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Breast feeding women.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product
* Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria number 8)
* Other malignancy within the last 5 years except: early stage cutaneous melanoma, adequately treated non-melanomatous skin cancer, curatively treated in situ cervical cancer, ductal carcinoma in situ (DCIS), FIGO Grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for >/= 5 years. Patients with a history of localised triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Absence of brain metastases is not required. Patients must not have symptomatic brain metastatic disease. The patient may be symptomatically controlled on a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
* Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of olaparib in combination with low dose thoracic radiotherapy | 1 year
Safety of olaparib in combination with low dose thoracic radiotherapy by evaluating participant toxicities and adverse events | 1 year
  For safety, all adverse events as determined by the investigator using CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Wu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Baptist Alliance Miami Cancer Institute, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org